CLINICAL TRIAL: NCT01005459
Title: Comparison of Spinal Tetracaine With Fentanyl and Epinephrine Versus Bupivacaine With Fentanyl and Epinephrine for Combined Spinal Epidural Labor Analgesia
Brief Title: Tetracaine Combined Spinal Epidural (CSE) Versus Bupivacaine CSE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: feasibility /drug availability issues - No study drug sources available
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB 9824
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-06

CONDITIONS: Labor Pain
Keywords: labor pain; combined spinal epidural labor analgesia; CSE analgesia; labor analgesia
MeSH Terms: conditions — Labor Pain | interventions — Tetracaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- tetracaine 2mg (Active Comparator)
  Interventions: Drug: Tetracaine
- Bupivacaine 2 mg (Active Comparator)
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Tetracaine — Tetracaine 2mg will be combined with Fentanyl 20 mcg and Epinephrine 50 mcg to treat labor pain.
  Arms: tetracaine 2mg
Drug: Bupivacaine — Bupivacaine 2 mg combined with fentanyl 20 mcg and Epinephrine 50 mcg will be used to treat labor pain.
  Arms: Bupivacaine 2 mg

SUMMARY:
The investigators hypothesis is that spinal tetracaine with fentanyl and epinephrine used for CSE labor analgesia volume will last a significantly longer period of time that that of spinal bupivacaine with fentanyl. After informed consent is obtained for the study, subjects meeting criteria when analgesia is requested will be randomized to receive a combined spinal-epidural containing either tetracaine 2 mg with fentanyl and epinephrine or bupivacaine 2 mg with fentanyl and epinephrine.

ELIGIBILITY:
Inclusion Criteria:

* early labor (>=2cm but =<6cm cervical dilation)
* at least 12 years of age
* have an assigned ASA physical status 1 or 2
* singleton pregnancy

Exclusion Criteria:

* contraindications to neuraxial anesthesia
* with allergies to drugs used in the study
* have an assigned ASA status 3 or 4
* advanced labor (> 6cm cervical dilation)
* less than 12 years of age
* Patients with the potential for distorted epidural anatomy, such as Harrington rods or prior back surgery, will also be excluded.

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-08; Primary Completion 2011-12-12 (Actual); Study Completion 2011-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter H. Pan, MD, Principal Investigator — WFUHS
Locations (1):
- Forsyth Medical Center- OB Anesthesia dept, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were approached after admission to the labor and delivery unit of our hospital about participation in this study
Period: Overall Study
Arm/Group | Tetracaine 2mg | Bupivacaine 2 mg
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tetracaine 2mg | Bupivacaine 2 mg | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 23 | 46
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 18 | 17 | 35
  african american | 5 | 2 | 7
  hispanic | 0 | 3 | 3
  other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Spinal Analgesic Duration
Description: duration of time in minutes from the time the combined spinal epidural is placed until the participant requests additional analgesia; at that time the epidural was dosed and study participation was complete
Time Frame: 1-2 hrs
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Tetracaine 2mg | Bupivacaine 2 mg
Number analyzed (Participants) | 23 | 23
minutes | 92.68 (46.71) | 89.61 (27.39)
Statistical Analysis 1: Comparison: Tetracaine 2mg; Test type: Other — unpaired t-test; p > 0.05, unpaired t-test compared between groups
Statistical Analysis 2: Comparison: Bupivacaine 2 mg; Test type: Other — unpaired t-test compared between groups; p > 0.05, unpaired t-test compared between groups

ADVERSE EVENTS:
Arm/Group | Tetracaine 2mg | Bupivacaine 2 mg
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes